CLINICAL TRIAL: NCT06536751
Title: Photobiomodulation in the Treatment of Spasticity in Children With Cerebral Palsy. A Controlled, Randomized, Blind Study
Brief Title: Therapeutic Photobiomodulation and Tretament of Spasticity
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Rebeca Boltes Cecatto, Professor M.D. Ph.D. Rebeca Boltes Cecatto, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CerebralPalsyPhotobio
Record Dates: First submitted 2024-07-19; First posted 2024-08-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Muscle Spasticity; Cerebral Palsy; Photobiomodulation; Low-Level Laser Therapy
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation (PBM) Treatment Group (Experimental): Photobiomodulation therapy sessions will be carried out in the physiotherapy environment on the University, once a week, for 08 consecutive weeks in the same day of the institution's standard physiotherapy session that the patient already uses regularly (not linked to the study). will be transcutaneously, punctual application of the LED in the medial and lateral gastrocnemius muscles of the right lower limb, in contact mode, 3J/cm2, with a 850nm wavelenght (01 point per gastroc, muscle). All patients will received the PBM protocol + the standard physiotherapy rehabilitation treatment of the institute not linked to the study, and which the patient already uses regularly.
  Interventions: Radiation: Photobiomodulation; Other: Institution's Standard Physiotherapy
- Photobiomodulation (PBM) Placebo Group (Placebo Comparator): PBM placebo therapy sessions will be carried out with the same characteristics of PBM treatment Group but with device turned off. All patients will received also the standard physiotherapy rehabilitation treatment of the institute not linked to the study, and which the patient already uses regularly.
  Interventions: Other: Institution's Standard Physiotherapy; Radiation: Photobiomodulation Placebo

INTERVENTIONS:
Radiation: Photobiomodulation — LED photobiomodulation therapy, once a week, for 08 consecutive weeks in the same day of the institution's standard physiotherapy session that the patient already uses regularly (not linked to the study). PBM will be transcutaneously, punctual application of the LED in the medial and lateral gastrocnemius muscles of the right lower limb, in contact mode, 3J/cm2, with a 850nm wavelenght.
  Other Names: Low Level Laser Therapy
  Arms: Photobiomodulation (PBM) Treatment Group
Other: Institution's Standard Physiotherapy — Physiotherapy treatment on the University, occur 2 therapeutic days per week, for 08 consecutive weeks (one of them in the same day of the PBM session). It consists of the use of motor physiotherapy, posture guidelines, stretching, positioning, joint range gain, ergonomics, sensory stimulation and proprioception, motor strengthening, tonus adjustment, functional training of upper and lower limbs, guidelines for the use of orthoses, stands, parapodium, parallel bars or wheelchair when needed. These are 45-minute sessions conducted by a physiotherapist.
  Other Names: Rehabilitation Physiotherapy
Radiation: Photobiomodulation Placebo — The same procedures of PBM group but device will be turned off
  Arms: Photobiomodulation (PBM) Placebo Group

SUMMARY:
Cerebral palsy is a non-progressive, permanent syndrome that occurs in childhood and is accompanied by motor, tônus and posture disorders. Its etiology is related to an insult or damage to the central nervous system in maturation. Approximately 80% of cerebral palsy course with spasticity, which, when left untreated, will generate pain and functional, anatomical and structural changes, with a negative impact. Photobiomodulation therapy has biological effects of tissue regeneration, muscle relaxation, vasodilation, reduction of the inflammatory process and relief of pain symptoms already described in the literature, in addition to being feasible, practical, safe, without side effects, painless and non-invasive.This study is a blind, randomized and controlled clinical trial that will evaluate the effect of photobiomodulation in reducing gastrocnemius muscle spasticity in children aged 2 to 18 years, diagnosed with spastic cerebral palsy of lower limbs of any etiology for at least 03 months and randomized into two groups: application of Low Intensity LED Therapy in the medial and right lateral gastrocnemius muscles (device power of 100mW, wavelength of 850nm, energy of 3J/cm2/point, once a week, making 08 therapeutic days during 02 months) or placebo group Low-Intensity LED Therapy (same device turned off). Both groups will also receive the standard treatment for spasticity. To assess the response to therapy, the outcomes evaluated will be the modified Ashworth Scale, the Mobility Domain of Pediatric evaluation of disability inventory, the Gross Motor Function Classification System scale and passive and active range of motion of the ankle analyzed at the pré and post each therapeutic session and in the pre and post therapeutic period of 08 sessions.

DETAILED DESCRIPTION:
Cerebral palsy is a non-progressive, permanent syndrome that occurs in childhood and is accompanied by motor, tonus and posture disorders. Its etiology is related to an insult or damage to the central nervous system in maturation, during the prenatal, perinatal or postnatal period, when the central nervous system has not yet fully developed.

Approximately 80% of cerebral palsy course with spasticity, which, when left untreated, will generate pain and functional, anatomical and structural changes in bones, joints, muscles, tendons and nerve junctions, with a negative impact on quality of life, social participation and functionality of this individual. In parallel, photobiomodulation therapy has biological effects of tissue regeneration, muscle relaxation, vasodilation, reduction of the inflammatory process and relief of pain symptoms already described in the literature, in addition to being feasible, practical, safe, without side effects, painless and non-invasive.Objectives and methods: this study is a pilot, double-blind, randomized and controlled clinical trial that will evaluate the effect of photobiomodulation in reducing gastrocnemius muscle spasticity in 28 children aged 2 to 18 years, diagnosed with spastic cerebral palsy of right lower limb of any etiology for at least 03 months, selected at the

Physiotherapy Service of Universidade Nove de Julho and randomized into two groups:

application of Low Intensity LED Therapy in the medial and right lateral gastrocnemius muscles (device power of 100mW, wavelength of 850nm, energy of 1.5 J/point, applied in 02 points per muscle, for 15 seconds, frequency of once a week, making 8 therapeutic days) or placebo group Low-Intensity LED Therapy (same device turned off). Patients with fixed anatomical deformity of the ankle with less than 90 degrees of dorsiflexion amplitude, malnutrition, severe gastroesophageal reflux disease and another type of associated movement disorder will be excluded. Both groups will also receive the standard treatment for spasticity performed by the hospital's rehabilitation health team.

To assess the response to therapy, the outcomes evaluated will be the modified Ashworth Scale (MAS), the Mobility Domain of Pediatric Evaluation of Disability Inventory for children (PEDI), the Gross Motor Function Classification System scale (GMFCS) and passive range of motion (ROM) of the ankle analyzed at the end of each therapeutic session and in the pre therapeutic period of 08 weeeks. Epidemiological data will be collected from the medical records of participants in the physiotherapy for characterizing the sample (age, gender,etiology of brain injury and type of paralysis, injury time, medications, comorbidities, previous surgeries, length of physiotherapy treatment at the start of the study, description of the physiotherapy treatment in use, use of a walking aid or orthosis. Data will be statistically analyzed and positive or negative results reported and discussed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of spastic cerebral palsy affecting inferior limbs from any etiology;
* Cerebral palsy duration at least 03 months;
* Patients ongoing physiotherapy treatment at University.

Exclusion Criteria:

* Patients with fixed anatomical deformities of the ankle that do not allow ankle joint movement of at least 90 degrees of amplitude;
* Patients with malnutrition;
* Patients who present acute clinical conditions with potential for increase spasticity such as acute fractures, skin ulcers, acute infections;
* Patients with severe gastroesophageal reflux disease;
* Patients with another type of movement or tone disorder;
* Patients who have exposed tumors in the area to be irradiated;
* Patients with a history of photosensitivity to photonic or light therapy;
* Patients who have undiagnosed lesions in the treatment region;
* Patients using topical photosensitizing medications or creams;

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 8 weeks (after PBM treatment) Spasticity Grade | At the basal assessment (baseline immediately before the PBM therapy), immediately after carrying out each session of PBM therapy, and 14 days after last session of PBM therapy
  Clinical evaluation of spasticity grade by Modified Asworth Scale (its performed by extending the patients limb first from a position of maximal possible flexion to maximal possible extension ( the point at which the first soft resistance is met). Afterwards, the modified Ashworth scale is assessed while moving from extension to flexion scoring
  0 No increase in tone
  1 slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension.
  1+ slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout ROM
  2 more marked increase in tone but more marked increased in muscle tone through most limb easily flexed
  3 considerable increase in tone, passive movement difficult
  4 limb rigid in flexion or extension

SECONDARY OUTCOMES:
Change from baseline to 8 weeks (after PBM treatment) Gross motor Classification System | At the basal assessment (baseline immediately before the PBM therapy), and 14 days after last session of PBM therapy
  Clinical evaluation with the aim of understanding the patient's situation in relation to their functional abilities and limitations
Change from baseline to 8 weeks (after PBM treatment) Passive range of motion of the ankle | At the basal assessment (baseline immediately before the PBM therapy), immediately after carrying out each session of PBM therapy, and 14 days after last session of PBM therapy
  Its measurement is carried out with the help of a goniometer. The measurement of passive ROM is done with a professional performing the movement through the evaluated
Change from baseline to 8 weeks (after PBM treatment) on mobility domain of Pediatric Evaluation of Disability Inventory | At the basal assessment (baseline immediately before the PBM therapy), and 14 days after last session of PBM therapy
  assesses key functional capabilities and performance in children ages 6 months to 7 years.

OTHER OUTCOMES:
Primary pilot statistical analysis | May 2025
  In an initial pilot evaluation checking safety trends, initial efficacy, or need for sample size adjustments, data from the first 12 participants that complete the intervention protocol, will be statistically analyzed (7 from PBM group and 5 from placebo group).

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca B Cecatto, Study Director — University of Nove de Julho; Ariane Zoll, Principal Investigator — Universiade Nove de Julho
Locations (2):
- Brazil (2):
  - Universidade Nove de Julho / Post-Graduate program Biophotonics Applied to Health Sciences, São Paulo, São Paulo
  - Universidade Nove de Julho / Post-Graduate program Biophotonics Applied to Health Sciences, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
The data will be share with Mendeley Data database or similar